CLINICAL TRIAL: NCT01815801
Title: Effect of Mechanical Ventilation on the Incidence of Pneumothorax After Subclavian Vein Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-1301-066-459
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Subclavian Vein Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ventilated group (Experimental): Lungs were mechanically ventilated during subclavian vein catheterization.
  Interventions: Other: Lungs were mechanically ventilated during subclavian vein catheterization
- Control group (Active Comparator): Lungs were not mechanically ventilated during subclavian vein catheterization.
  Interventions: Other: Lungs were not mechanically ventilated during subclavian vein catheterization

INTERVENTIONS:
Other: Lungs were not mechanically ventilated during subclavian vein catheterization — Control group
  Arms: Control group
Other: Lungs were mechanically ventilated during subclavian vein catheterization — Ventilated group
  Arms: Ventilated group

SUMMARY:
The purpose of this study is to determine whether mechanical ventilation influences the incidence of pneumothorax after subclavian venous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing neurosurgery that requires the placement of subclavian venous catheterization

Exclusion Criteria:

* infection over the puncture site
* history of prior clavicular fracture
* anatomical anomaly of subclavian vein
* Pneumothorax

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
incidence of pneumothorax | an expected average of one day after surgery
  Postoperative chest X-ray will be taken to check for the occurence of pneumothorax.

SECONDARY OUTCOMES:
catheterization success rate | an expected average of one day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea